CLINICAL TRIAL: NCT02693821
Title: Persistent Postoperative Pain Incidence With Long Term Perioperative Gabapentin Used
Brief Title: Persistent Postoperative Pain Incidence With Gabapentin Used
Acronym: PPP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, FRANCISCO CARLOS BONOFIGLIO, Anesthesiology Doctor, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2575
Record Dates: First submitted 2016-02-19; First posted 2016-02-29 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Pain, Postoperative
Keywords: Gabapentin; prevention; incidence
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: Estudio Controlado, randomizado, prospectivo y ciego.
Who Masked: Participant, Investigator
Masking Description: Cuando el paciente dé su consentimiento, será reclutado y randomizado a un grupo control (recibirá placebo) o a un grupo tratamiento (recibirá gabapentin) Los pacientes recibirán una técnica anestésica habitual, basadas en drogas endovenosas mediante el método TCI (target controlled infusión). Con este método se unifica el uso de las drogas anestésicas, que son utilizadas de acuerdo a sexo, edad, género, peso y altura en cada uno de los pacientes.
  La analgesia será la convencional para cada cirugía y se continuará con el uso de catéteres epidurales, para analgesia en aquellas intervenciones donde su aplicación sea habitual.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gabapentin (Experimental): 300mg of Gabapentin per day (two doses), orally during 30 days
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): 300mg of Placebo per day (two doses), orally during 30 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Gabapentin — gabapentin 300 mg per day, orally during 30 days
  Arms: Gabapentin
Drug: Placebo — Placebo 300 mg per day, orally during 30 days
  Arms: Placebo

SUMMARY:
The study's objective will be to evaluate the gabapentine efficiency in orally and long term used after painfully surgeries.

DETAILED DESCRIPTION:
This study will be: controlled, prospective, randomized and double blind.

Its main objective will be to evaluate the pre and postoperative Gabapentin efficiency in orally doses and long term used of it in order to prevent or decrease persistent postoperative pain (PPP) in surgeries with high incidence of it (Pain). Patients will be randomly divided in two branches; one of them will take 600 mg of Gabapentin twice a day and the other group will take Placebo (twice a day also).

Both groups of patients will have to take one pill the day before the surgery (300 mg) and other pill on the surgery day (300mg). After that, the patients will have to continue this treatment during 30 days (two doses per day of Gabapentin or placebo).

After the surgery and after taking the second pill, it will be evaluated:

postoperative sharp pain, sickness, vomiting, sedation and adverse effects.

Patients will be evaluated in the pain treatment office (consulting room) the following times:

1. 30 days after the surgery. (taking drugs suspended)
2. 3 month after the surgery.
3. 6 months after the surgery.
4. 12 months after the surgery

This monitoring treatment will be done in order to evaluate the presence or absence of persistent postoperative pain (PPP).

ELIGIBILITY:
Inclusion Criteria:

* Patients that require persistent painfully surgeries such as breast surgeries (mastectomies and breast implants), herniorrhaphies (not laparoscopical) unilateral or bilateral, amputations of upper and lower limbs and chest surgeries (thoracotomy, thoracoscopy , sternotomies).
* Patients that had already signed the informed consent.
* Patients aged between 21 and 75.
* ASA I - II _ III (Classification system that the American Society of Anesthesiologists (ASA) uses to estimate the anesthesiology risk that patients may suffer)
* BMI, not more than 35 Kg/m2.

Exclusion Criteria:

* Pregnant women
* Patients that suffer liver and renal failure (plasma creatinine over 1.5 mg/ml or creatinine clearance less than 60 ml/min),heart failure or neurological dysfunction.
* Diabetic patients
* Gabapentine allergic patients

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2015-12; Primary Completion 2016-01 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of pain after using gabapentin. | Two years
  It will be used a 10cm ruler which will allows the patients indicates how much pain they are feeling at the moment, where 0 is no pain at all and 10 is the maximum imaginable pain.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco FB Bonofiglio, Doctor, Study Director — Hospital Italiano de Buenos Aires
Locations (1):
- Sofía Konekny, Almagro, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Macrae WA. Chronic post-surgical pain: 10 years on. Br J Anaesth. 2008 Jul;101(1):77-86. doi: 10.1093/bja/aen099. Epub 2008 Apr 22. PMID 18434337
- [Background] Werner MU, Kongsgaard UE. I. Defining persistent post-surgical pain: is an update required? Br J Anaesth. 2014 Jul;113(1):1-4. doi: 10.1093/bja/aeu012. Epub 2014 Feb 18. No abstract available. PMID 24554546
- [Background] Borsook D, Kussman BD, George E, Becerra LR, Burke DW. Surgically induced neuropathic pain: understanding the perioperative process. Ann Surg. 2013 Mar;257(3):403-12. doi: 10.1097/SLA.0b013e3182701a7b. PMID 23059501
- [Background] Crombie IK, Davies HT, Macrae WA. Cut and thrust: antecedent surgery and trauma among patients attending a chronic pain clinic. Pain. 1998 May;76(1-2):167-71. PMID 9696470
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Gilron I, Watson CP, Cahill CM, Moulin DE. Neuropathic pain: a practical guide for the clinician. CMAJ. 2006 Aug 1;175(3):265-75. doi: 10.1503/cmaj.060146. PMID 16880448
- [Background] Matthews EA, Dickenson AH. Effects of spinally delivered N- and P-type voltage-dependent calcium channel antagonists on dorsal horn neuronal responses in a rat model of neuropathy. Pain. 2001 May;92(1-2):235-46. doi: 10.1016/s0304-3959(01)00255-x. PMID 11323145
- [Background] Schmader KE. Epidemiology and impact on quality of life of postherpetic neuralgia and painful diabetic neuropathy. Clin J Pain. 2002 Nov-Dec;18(6):350-4. doi: 10.1097/00002508-200211000-00002. PMID 12441828
- [Background] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Background] Backonja MM, Galer BS. Pain assessment and evaluation of patients who have neuropathic pain. Neurol Clin. 1998 Nov;16(4):775-90. doi: 10.1016/s0733-8619(05)70097-9. PMID 9767062
- [Background] Lavand'homme P. From preemptive to preventive analgesia: time to reconsider the role of perioperative peripheral nerve blocks? Reg Anesth Pain Med. 2011 Jan-Feb;36(1):4-6. doi: 10.1097/AAP.0b013e31820305b8. No abstract available. PMID 21455081
- [Background] Rosner H, Rubin L, Kestenbaum A. Gabapentin adjunctive therapy in neuropathic pain states. Clin J Pain. 1996 Mar;12(1):56-8. doi: 10.1097/00002508-199603000-00010. PMID 8722736
- [Background] Dauri M, Faria S, Gatti A, Celidonio L, Carpenedo R, Sabato AF. Gabapentin and pregabalin for the acute post-operative pain management. A systematic-narrative review of the recent clinical evidences. Curr Drug Targets. 2009 Aug;10(8):716-33. doi: 10.2174/138945009788982513. PMID 19702520
- [Background] Miller A, Price G. Gabapentin toxicity in renal failure: the importance of dose adjustment. Pain Med. 2009 Jan;10(1):190-2. doi: 10.1111/j.1526-4637.2008.00492.x. Epub 2008 Aug 18. PMID 18721173